CLINICAL TRIAL: NCT00861952
Title: The Safety and Efficacy of Neuragen in Diabetic Peripheral Neuropathy: A Double-blind Randomized Placebo Controlled Trial
Brief Title: Neuragen for Peripheral Diabetic Neuropathy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study has received ethics approval, however funding limitations have resulted in suspending date of commencement.
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Kieran Cooley, Associate Director, Research, The Canadian College of Naturopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCNM-0901
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Diabetic Peripheral Neuropathy; Diabetic Neuralgia
Keywords: Diabetic peripheral neuropathies; Neuralgia; Complementary medicine; Analgesia
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia; Agnosia | interventions — Mineral Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neuragen (Experimental): Ad lib use of Neuragen (a natural health product) applied topically 2-3 times per day in 2-3 drops per application
  Interventions: Other: Neuragen
- Mineral oil (Sham Comparator): Mineral oil, scent and color matched to intervention
  Interventions: Other: Mineral oil

INTERVENTIONS:
Other: Neuragen — 2-3 drops applied topically 2-3 times per day as needed over a 3 month period
  Arms: Neuragen
Other: Mineral oil — Ad lib use of mineral (scent and color matched to Neuragen) applied topically 2-3 times per day in 2-3 drops per application
  Arms: Mineral oil

SUMMARY:
The purpose of this study is to determine if the use of Neuragen (a natural health product oil rubbed into the skin) is effective at reducing pain and improving the quality of life in people with diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Incidence of diabetic neuropathy and development of diabetic ulcers varies based on the severity (lack of blood sugar control) and duration of diabetes. Estimates of rates of occurrence vary although one prospective study showed 7.2% of newly diagnosed ulcer-free diabetics developed ulcers within one year of being diagnosed. Current treatment initiatives aimed at educating diabetic patients on how to prevent diabetic ulcers and mange peripheral neuropathy have had varied success. Chronic pain is the number one reason that this population seeks help from medical professionals. Diabetics are particularly predisposed to a potentially disabling form of chronic pain known as peripheral neuropathy. In fact, over 50% of diabetics have painful neuropathy, or will develop this condition. Other than the primary goal of addressing blood sugar levels, conventional treatment of diabetic peripheral neuropathy involves prescription gabapentanoids or opiod analgesics, both of which have considerable cost and may be associated with side effects from long-term use and overall limited success rates. Neuragen is an over-the-counter natural health product that may be a safe and effective treatment option for this disease. Using a randomized double-blind placebo control clinical trial the effects of Neuragen on pain, function and quality of life will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of at least 18 years of age
* Established diagnosis of neuropathic pain for at least the past 3 months duration, and type 1 or type 2 diabetes, confirmed by primary care physician and/or neurologist. By signing the informed consent, participants agree to have the study coordinator contact their physician for confirmation of diagnosis.
* Pain of at least level 4 on a 0-10 scale, and not over 9, despite other treatments on intake.
* Presence of dynamic tactile allodynia or pinprick hyperalgesia
* Normal cognitive and communication skills (as judged by investigator) and ability to complete self-report questionnaires.

Exclusion Criteria:

* Pregnancy
* Previous or continuing use of Neuragen®
* Evidence of other types of pain as, or more severe, than the pain under study
* Major psychological conditions requiring treatment
* History of eczema/atopy/anaphylaxis or unusual skin reactions. This will be assessed using a subjective question (Have you ever suffered from eczema? Or experienced a skin reaction to a substance? Or experienced an anaphylactic reaction?)
* Self reported sensitivity to perfumes, essential oils, odors.
* Changes to current pain management regime within the previous month prior to start of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01

PRIMARY OUTCOMES:
Brief Pain Inventory for sustained relief | Baseline to month 3
Numeric pain scale (0-10) for immediate relief | Baseline compared to average daily measure over 3 months

SECONDARY OUTCOMES:
NeuroQol-97 quality of life measurement questionnaire | Baseline to 3 months
Liver enzyme - AST | Baseline to 3 months
Liver enzyme - ALT | Baseline to 3 months
Liver enzyme - GGT | Baseline to 3 months
Neurologic impairment scale LL +7 | Baseline to 3 months
Amount of medication used | Baseline to 3 months
Adverse event reports | Baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lynch, MD, Study Chair — Dalhousie University; Kieran Cooley, ND, Principal Investigator — The Canadian College of Naturopathic Medicine
Locations (2):
- Canada (2):
  - Pain Management Unit, Halifax, Nova Scotia
  - Robert Schad Naturopathic Clinic, Toronto, Ontario